CLINICAL TRIAL: NCT07164222
Title: Triglycerides Glucose Index on Diabetic Patients Type 2
Brief Title: Triglycerides Glucose Index and Ratio on Diabetic Type 2
Acronym: Diabetes 2
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, DEAAELDIN MOHAMED SEDEK, Consultant of Internal Medecine, Assiut University
Other Study IDs: Triglycerides .glucose index
Record Dates: First submitted 2025-09-02; First posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Triglycerides Glucose Index and Ratio on Diabetic Type 2

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Age between 18years and 65years old with studies of complications of diabetes type 2 with high index: Clinical and laboratory follow up complications of diabetes with high triglycerides glucose index and ratio
  Interventions: Diagnostic Test: Glycated haemoglobin and triglycerides level

INTERVENTIONS:
Diagnostic Test: Glycated haemoglobin and triglycerides level — Follow up with triglycerides and glucose index and ratio on diabetic type 2

SUMMARY:
Triglycerides glucose index and ratio on diabetic type 2

DETAILED DESCRIPTION:
Triglycerides glucose index and ratio on patients with type 2 diabetes mellitus and microvacular complications

ELIGIBILITY:
Inclusion Criteria:

* above 18years under 65years

Exclusion Criteria:

Type 1 diabetic Under 18years Severe complications Icu patients Blind and handicapped patients

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Triglycerides glucose index and ratio on diabetic type 2
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-09-30 (Estimated); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Follow up with routine investigations for diabetic cases | 2years
  Microvacular complications with diabetic

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Ali Obedollah, MD, Study Director — Faculty of science, Assiut university

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Khalaji A, Behnoush AH, Khanmohammadi S, Ghanbari Mardasi K, Sharifkashani S, Sahebkar A, Vinciguerra C, Cannavo A. Triglyceride-glucose index and heart failure: a systematic review and meta-analysis. Cardiovasc Diabetol. 2023 Sep 7;22(1):244. doi: 10.1186/s12933-023-01973-7. PMID 37679763
- [Background] dmsjournal.biomecentral.com
- See also: Related Info — https://Pubmed.ncbi.nlm.nih.gov